CLINICAL TRIAL: NCT04377425
Title: COVID-19 Prevalence, Morbidity and Long Term Cognitive Deficits in Consecutive Patients Presenting With Acute Neurological Symptoms
Brief Title: COVID-19 Prevalence and Cognitive Deficits in Neurological Patients
Acronym: Neuro-Covid
Status: Withdrawn | Type: Observational
Why Stopped: No acute neurological patients presented with concomitant COVID-19
Sponsor: Aarhus University Hospital (Other)
Responsible Party: Principal Investigator, Grethe Andersen, Professor, DMSc, senior consultant, Aarhus University Hospital
Other Study IDs: Neuro-Covid-19
Record Dates: First submitted 2020-04-29; First posted 2020-05-06 (Actual); Last update posted 2020-09-03 (Actual); Status verified 2020-09

CONDITIONS: Neurological Diseases or Conditions; Stroke, Acute; Seizure Disorder
Keywords: COVID-19; Neurological disease; Prevalence; Cognitive outcome; Stroke; Seizure/epilepsy
MeSH Terms: conditions — Stroke; Epilepsy; COVID-19; Nervous System Diseases; Seizures

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — For study participants in the extended study:
  Blood samples (13mL) and cerebrospinal fluid (7mL) will be collected at baseline
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Patients with acute neurological symptoms: Consecutive patients with acute neurological disease admitted at the Neurology departments will be tested with a nasopharyngeal swap for SARS-COVID-19 RNA according to standard operating procedures at the department (if estimated hospital stay is >24hours). Medical and clinical characteristics will be collected
  Interventions: Diagnostic Test: COVID-19 swap test PCR
- Stroke patients: COVID-19 positive patients will be asked to participate in the extended study together with matched COVID-19 negative controls.
  Extended study: Collection of cerebrospinal fluid and blood-samples, clinical and cognitive assessment at baseline and at 3-month follow-up
  Interventions: Diagnostic Test: COVID-19 swap test PCR
- Seizure/epilepsy: COVID-19 positive patients will be asked to participate in the extended study together with matched COVID-19 negative controls.
  Extended study: Collection of cerebrospinal fluid and blood-samples, clinical and cognitive assessment at baseline and at 3-month follow-up
  Interventions: Diagnostic Test: COVID-19 swap test PCR

INTERVENTIONS:
Diagnostic Test: COVID-19 swap test PCR — COVID-19 swap test PCR performed according to hospital standard operating procedures

SUMMARY:
The purpose is to investigate the COVID-19 prevalence, associated morbidity and long-term cognitive deficits in consecutive patients presenting with acute neurological symptoms

DETAILED DESCRIPTION:
Severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2), is spreading in nearly every country in the world. Patients with coronavirus disease 2019 (COVID-19) typically present with cough, fever and respiratory illness. In another coronavirus (SARS-COV-1) causing the SARS outbreak in 2002 to 2003, neurons have been found to be highly susceptible for infection and the virus can cause extensive neuronal damage with only minimal respiratory affection. Similar to SARS-CoV-1, COVID-19 virus exploits the angiotensin-converting enzyme 2 (ACE-2) receptor to gain entry and infect cells. Both glial and neurons express ACE-2 receptors and makes them potential targets, however the neurotropic potential in humans remain largely undescribed. Neurological manifestations of COVID-19 have only been sporadically described in single or short series of case reports together with a case of COVID-19 RNA in the cerebrospinal fluid.

Loss of smell (anosmia) may be a presenting symptom in COVID-19. Interestingly, in a study from Italy anosmia was present in 19,4% and not typical accompanied by nasal obstruction, rhinitis or sinusitis, making direct damage and invasion of the olfactory nerve more likely. A Chinese study have found that 36.6% of COVID-19 patients experience neurological symptoms and that severely affected COVID-19 patients reported more neurological symptoms.

In general, neurological manifestations to viral disease may occur as a direct result of viral invasion and damage to either the central or peripheral nervous system or from an immune mediated neurological damage either during (para) or after (post) the viral infection. Furthermore, the inflammation in itself can increase the risk of arterial thrombosis and thus ischemic stroke.

Early reports from Italy stresses the need to pay attention to neurological symptoms, as they are often neglected due to the systemic and respiratory impairment. Further, concerning reports from the Center for Disease Control (CDC) in USA, have estimated that out of COVID-19pos patients up to 46.5% may be asymptomatic/pre-symptomatic and 17,5% never develop classical COVID-19 symptoms. The COVID-19 infection is likely to be missed if patients present with symptoms from another organ system. Moreover, it poses a transmission risk for other admitted patients and healthcare workers and a risk that a possible association between e.g. neurological symptoms/diseases and a COVID-19 infection are missed. The role and presence of COVID-19 infection in patients presenting with acute neurological symptoms is currently unknown.

ELIGIBILITY:
Eligibility criteria for the extended study:

Inclusion Criteria:

* Adult patients
* New onset of neurological symptoms
* Independent in daily activities (modified Rankin Scale ≤ 2)
* Stroke or epilepsy/seizure

Exclusion Criteria:

* Pre-existing neurodegenerative disease
* Diagnosed with cerebral neoplasm
* Pre-existing expected life expectancy < 3 months
* Suspected non-organic (functional) disorder

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Base study: Consecutive patients with acute neurological disease admitted at the Neurology department at Aarhus University Hospital will be tested with a nasopharyngeal swap for SARS-COVID-19 RNA
  Extended study: Patients fulfilling the extended study criteria will be asked to participate in extended study depending on their COVID-19 status and whether study criteria are fulfilled
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-05-07 (Estimated); Primary Completion 2020-11-29 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of COVID-19 infection in consecutive patients with neurological symptoms | 6 months
  To investigate the prevalence of COVID-19 infections in consecutive patients with acute onset of neurological symptoms (with or without prior neurological disease)

SECONDARY OUTCOMES:
Three months cognitive function of COVID-19 positive patients | 3 months
  Three months cognitive function (Montreal Cognitive Assessment) of COVID-19 positive patients compared to COVID-19 negative patients
Clinical presentation of neurological symptoms in COVID-19 positive patients | 6 months
  Characterization of the neurological symptoms in neurological COVID-19 positive patients (exploratory endpoint)
Prevalence of pre- and asymptomatic COVID-19 positive patients in acutely admitted neurological patients | 6 months
  Prevalence of pre-symptomatic and asymptomatic COVID-19pos in acutely admitted patients with a primary complaint of neurological symptoms.
Anosmia in COVID-19 positive patients | 6 months
  Prevalence of anosmia in COVID-19pos patients compared to COVID-19neg patients
Exploratory analysis on neuro-specific and inflammatory blood and cerebrospinal fluid markers of COVID-19 infection | 24 months
  Neuro-specific and inflammatory blood- and cerebrospinal fluid markers in COVID-19 positive patients compared to COVID-19 negative matched controls
Exploratory analysis of the coagulation profile of COVID-19 positive patients compared to COVID-19neg patients | 24 months
  Functional and immunologic plasma assays will be employed to analyze proteins and pathways in coagulation and fibrinolysis

CONTACTS AND LOCATIONS:
Overall Officials: Grethe Andersen, MD, Principal Investigator — Aarhus University Hospital
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Aalborg, DK
  - Aarhus University Hospital, Aarhus, DK
  - Regional Hospital West Jutland, Hostebro, Holstebro, DK
  - Regional Hospital Central Jutland, Viborg, Viborg, DK

IPD SHARING:
Plan to Share IPD: Undecided
Upon reasonable request